CLINICAL TRIAL: NCT07190053
Title: Long-term Treatment Strategies and Effectiveness of Secukinumab in Juvenile Idiopathic Arthritis Patients of Psoriatic and Enthesitis-related Arthritis Categories: Secondary Use of Data and Primary Data Collection From the German BIKER Registry
Brief Title: Long Term Treatment Strategies and Effectiveness of Secukinumab in Patient With JIA Subtypes of JPsA and ERA: Study From German BIKER Registry.
Status: Not yet recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457V12401
Record Dates: First submitted 2025-06-12; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Enthesitis-related Arthritis (ERA); Juvenile Psoriatic Arthritis (JPsA)
Keywords: ERA,; JPsA,; secukinumab
MeSH Terms: conditions — Arthritis, Juvenile | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Secukinumab: All children and adolescents with ERA or JPsA who received at least one dose of secukinumab.
  Interventions: Other: Secukinumab

INTERVENTIONS:
Other: Secukinumab — This is an observational study, there is no treatment allocation

SUMMARY:
The goal of this study is to understand the long-term treatment strategies in children and adolescents diagnosed with ERA or JPsA who received secukinumab and achieved inactive disease and to evaluate the long-term treatment effectiveness of secukinumab in the ERA or JPsA patients in the postauthorization setting.

DETAILED DESCRIPTION:
This is a multicenter, non-interventional cohort study with a combined data collection principle based on secondary use of data and primary data collection from the existing BIKER registry among pediatric patients with a recorded diagnosis of ERA or JPsA who have been treated with secukinumab.

The primary objective of this study is to characterize potentially less demanding long-term treatment strategies (e.g., dose tapering, treatment withdrawal followed by treatment re-initiation as needed) and to characterize their effectiveness (evaluated by occurrence of disease flares) in children and adolescents with Enthesitis-Related Arthritis (ERA) or Juvenile Psoriatic Arthritis (JPsA) categories documented in the German Biologics in pediatric rheumatology (BIKER) registry who received secukinumab and achieved inactive disease.

The date of first treatment/prescription of secukinumab will be considered as the index date. The baseline period to evaluate the demographic and clinical characteristics includes the index date and up to 1 year prior to the index date; if no record is available at the index date whichever record is closest to the index date will be used. For JIA-related variables, such as JIA-related manifestations, the evaluation will not have a specific time limit prior to the index date."

ELIGIBILITY:
Inclusion Criteria:

* In the BIKER registry, males and females ≥ 6 years old and ≤ 17 years old diagnosed with ERA according to the ILAR-criteria or JPsA according to the ILAR or the Vancouver criteria, who initiated at least one dose of secukinumab after it was approved in Germany and according to the label.
* Written informed consent from parent/legal guardian and assent from minor patient (11-17 years of age) for participating in the BIKER registry and for this study enrolment.

Exclusion Criteria:

* Patients taking other biologic immunomodulating agent(s) or Janus kinase (JAK) inhibitors concomitantly with secukinumab at index date.
* Patients participating in any interventional trials at index date.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents diagnosed with ERA or JPsA JIA categories who received secukinumab
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-09-18 (Estimated); Study Completion 2029-09-18 (Estimated)

PRIMARY OUTCOMES:
Number of patients who had the following long-term treatment strategy after achieving inactive disease on secukinumab | Up to 5 years
  Number of patients who had the following long-term treatment strategy after achieving inactive disease on secukinumab
  * Secukinumab treatment remained unchanged or dose was increased.
  * Dose tapering of secukinumab (by dose reduction or prolongation of treatment interval).
  * Increase of secukinumab dose after a tapering period.
  * Initiation of other biologics after a tapering period.
  * Entering a secukinumab-free period due to achieving inactive disease or clinical remission (stratified by those who discontinue secukinumab due to achieving inactive disease without achieving clinical remission and those who achieve clinical remission)
  * Re-initiation of secukinumab after a secukinumab-free period
  * Initiation of other biologics after a secukinumab-free period
Number of patients experiencing at least one episode of flare | Up to 5 years
  Number of patients experiencing at least one episode of flare:
  * Following inactive disease for patients whose secukinumab treatment remained unchanged or increased dose.
  * Following the start of tapering or discontinuation of secukinumab treatment after achieving inactive disease

SECONDARY OUTCOMES:
Number of patients with following secukinumab treatment patterns | every 3 months after index date until end of follow-up, up to 5 years
  Number of patients with following secukinumab treatment patterns:
  * Secukinumab treatment remained unchanged or dose was increased
  * Dose tapering of secukinumab (by dose reduction or prolongation of dosing interval)
  * Increase of secukinumab dose after a tapering period.
  * Initiation of other biologics after a tapering period.
  * Discontinuation of secukinumab:
  * Switching directly from secukinumab to other therapies.
  * Entering a secukinumab-free period.
  * Re-initiation of secukinumab after a secukinumab-free period.
  * Initiation of other biologics after a secukinumab-free period.
Number of participants by reason for changes to treatment strategy | every 3 months after index date until end of follow-up, up to 5 years
  The reason for changes to treatment strategy:
  * Achieving inactive disease
  * Achieving clinical remission
  * Lack of effectiveness
  * Occurrence of adverse events
  * Patient's /Parent's decision
  * Other
Number of patients achieving Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 30/50/70/90 criteria at follow-up | Every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  The adapted ACR Pediatric 30/50/70/90 criteria was used to determine efficacy defined as improvement from baseline of at least 30/50/70/90% respectively in at least 3 of the following 6 components
  * Physician's Global Assessment of disease activity on a 0-100 mm VAS from 0 mm = no disease activity to 100 mm = very severe disease activity.
  * Parent's or patient's Global Assessment of Subject's overall wellbeing on a 0-100 mm VAS from 0 mm= very well to 100 mm= very poor.
  * Functional ability: Childhood Health Assessment Questionnaire (CHAQ©)
  * Number of joints with active arthritis using the ACR definition (The ACR definition of active arthritis is any joint with swelling, or in the absence of swelling, limitation of motion accompanied by either pain on motion or tenderness not due to deformity)
  * Number of joints with limitation of motion
  * Laboratory measure of inflammation: CRP (mg/L)
Number of patients achieving at least minimal disease activity | Every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  Patients who achieved minimal disease activity and inactive disease can be defined based on JADAS-10 score. JADAS-10 is a composite disease activity score for JIA including four measures:
  * physician's global assessment of disease activity (NRS)
  * parent/guardian's or patient's global assessment of overall wellbeing (NRS)
  * number of joints (up to 10) with active arthritis
  * CRP/ESR, whichever is available
Number of patients achieving inactive disease | Every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  Inactive disease is achieved if either of the following two criteria is fulfilled:
  * Wallace et al (2011) ACR criteria for inactive disease:
  * no joints with active arthritis
  * no active uveitis
  * normal CRP/ESR, or if elevated, not attributable to JIA
  * physician's global assessment of disease activity ≤ 1 (NRS)
  * duration of morning stiffness attributable to JIA ≤ 15 minutes
  * JADAS-10 score-based definition for inactive disease:
  * physician's global assessment of disease activity (NRS)
  * parent/guardian's or patient's global assessment of overall wellbeing (NRS)
  * number of joints (up to 10) with active arthritis
  * CRP/ESR, whichever is available
Number of patients achieving clinical remission | Every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  Patients with 6 consecutive months of inactive disease are defined as entering clinical remission.
Number of patients achieving complete resolution of dactylitis and enthesitis. | Every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  Number of patients achieving complete resolution of dactylitis and enthesitis.
Change from baseline in pain score | Every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  Change from baseline in pain score through numeric rating scale (NRS). Numeric rating scale spans from 0 (no pain) to 10 (strongest pain).
Change from baseline in JIA ACR criteria individual components | Every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  Summary of JIA ACR core components for all subjects and each JIA category.
  Negative percent change indicates improvement.
  JIA ACR criteria individual components:
  * Number of joints with active arthritis
  * Number of joints with limited range of motion
  * C-reactive protein (CRP) or erythrocyte sedimentation rate (ESR), whichever is available.
  * Functional status using the Childhood Health Assessment Questionnaire (CHAQ) disability index and Health Assessment Questionnaire for adults.
  * Physician global assessment of overall well-being through NRS.
  * Parent/guardian's or patient's global assessment of overall well-being through NRS.
Change from baseline in JADAS-10 individual criteria: | Baseline, up to 5 years
  JADAS-10 stands for Juvenile Arthritis Disease Activity Score, with up to 10 joints assessed for active arthritis as part of the score. JADAS-10 individual criteria are:
  * Physician's global assessment: NRS scale - 0 (inactive disease ) to 10 (active disease)
  * Parent/guardian's or patient's global assessment: NRS scale - 0 (inactive disease ) to 10 (active disease)
  * Number of joints with active arthritis: from 0 active joints to 10 active joints.
  * CRP/ESR, whichever is available: Westergren erythrocyte sedimentation rate (ESR), normalized to a 0-10 scale. The CRP was truncated to a 0-10 scale accord¬ing to the following formula: (CRP (mg/l)-10)/10, similar to the normalized ESR used in the original JADAS.
  Before calculation, CRP values <10 mg/l were converted to 10 and CRP values >110 mg/l were converted to 110.
JADAS-10 score | At baseline and every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  JADAS-10 stands for Juvenile Arthritis Disease Activity Score, with up to 10 joints assessed for active arthritis as part of the score. The score spans from 0 to 40. Lower values mean lower activity and higher values mean higher activity.
Change from baseline in swollen joint count | Every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  Change from baseline in swollen joint count
Change from baseline in tender joint count | Every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  Change from baseline in tender joint count
Total dactylitis count | At baseline and every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  Total dactylitis count
Total enthesitis count | At baseline and every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  Total enthesitis count, number of affected sites.
Enthesitis score | At baseline and every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  The Enthesitis score using Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) asks for evaluation of swelling and tenderness at different anatomical locations.
  All locations are scored as 0 "no activity" or 1 "activity". The MASES is the sum of all site scores.
Number of participants by JIA-related manifestations | At baseline and every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  JIA-related manifestations:
  * Uveitis presence.
  * Serositis presence.
  * General lymphadenopathy presence.
  * Fever presence.
Modified Schoeber's test to assess axial mobility (ERA only). | At baseline and every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  Modified Schober's test is measuring lumbar spine mobility quantitatively. It measures lumbar spine flexion range of motion.
  To conduct the test, the patient stands upright. The examiner locates the two posterior superior iliac spines and draws a horizontal line between them. A second point is marked 15cm above this line.Then the patient is asked to bend forwards as far as possible whilst keeping the knees fully extended. The distance between the previously marked points is measured again and indicates the amount of flexion.
Overall and nocturnal back pain NRS (ERA only). | At baseline and every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  For patients with Enthesitis-Related Arthritis (ERA), the overall and nocturnal back pain through NRS will be recorded. NRS stands for Numerical Rating Scale: 0 (no pain) to 10 (strongest pain).
Skin involvement using the Investigator Global Assessment Modified (IGA Mod) 2011 score (JPsA only). | At baseline and every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  The IGA Mod is a simple score for the evaluation of psoriasis:
  0 = clear (e.g., no signs of psoriasis, some post-inflammatory hyperpigmentation may be present);
  1. = almost clear (e.g., no thickening, normal or pink coloration);
  2. = mild (e.g., mild thickening, pink to light red coloration),
  3. = moderate (e.g., moderate thickening, dull to bright red);
  4. = severe (e.g., severe thickening, bright to deep red).
Psoriasis Area Severity Index (PASI) (JPsA only). | At baseline and every 3 months after index date until the end of follow-up or until secukinumab discontinuation or switching to another biologic, whichever occurs first, up to 5 years
  For patients with Juvenile Psoriatic Arthritis (JPsA), the PASI score will be calculated. The PASI is used for assessing and grading the severity of psoriatic lesions and their response to therapy. PASI scores can range from a lower value of 0, corresponding to no signs of psoriasis, up to a theoretic maximum of 72.0.
Number of participants with relevant JIA-related manifestations | Baseline
  Number of patients with relevant Juvenile Idiopathic Arthritis (JIA)-related manifestations (such as uveitis, serositis)
Time from symptom onset to diagnosis of ERA or JPsA | Baseline
  Time from symptom onset to diagnosis of Enthesitis-Related Arthritis (ERA) or Juvenile Psoriatic Arthritis (JPsA)
Disease duration at the time of secukinumab initiation | Baseline
  Disease duration at the time of secukinumab initiation
Therapy duration prior to start of secukinumab | Baseline
  Therapy duration prior to start of secukinumab (including all drug and non-drug therapies prescribed for ERA or JPsA)
Number of treatment lines prior to start of secukinumab | Baseline
  Number of treatment lines prior to start of secukinumab
Prior medication | Baseline
  Prior medication and dosage (including all drug and non-drug therapies prescribed for ERA or JPsA)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com